CLINICAL TRIAL: NCT02087423
Title: A Phase II,Non-comparative,Open Label, Multi-centre, International Study of MEDI4736, in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer (Stage IIIB-IV) Who Have Received at Least 2 Prior Systemic Treatment Regimens Including 1 Platinum-based Chemotherapy Regimen
Brief Title: A Global Study to Assess the Effects of MEDI4736 (Durvalumab) in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer
Acronym: ATLANTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4191C00003; 2013-005427-16 (EudraCT Number)
Record Dates: First submitted 2014-03-04; First posted 2014-03-14 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Locally advanced, metastatic, Non-Small Cell Lung Cancer, MEDI4736, Durvalumab, PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- MEDI4736 (Experimental): see below
  Interventions: Drug: MEDI4736

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 (durvalumab) by intravenous infusion every two weeks. Treatment from Day 1 for a maximum of 12 months or study drug withdrawal if this occurs earlier. Patients who achieve CR, PR or SD through the end of the initial 12-month treatment period can restart treatment with MEDI4736 (durvalumab) when they eventually do progress. This retreatment period can continue for as long as the investigator considers to patient to be receiving clinical benefit.

SUMMARY:
A study to assess the Effects of MEDI4736 (Durvalumab) in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer in terms of efficacy, safety and tolerability

DETAILED DESCRIPTION:
This study is designed to investigate the efficacy, safety, tolerability of a new drug, MEDI4736 (Durvalumab), in patients with Locally Advanced or Metastatic Non Small Cell Lung Cancer. MEDI4736 will be investigated in patients who have received at least two prior treatment regimens including one platinum-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years.
* Documented evidence of NSCLC (stage IIIB/IV disease)
* Disease progression or recurrence after both a platinum-based chemotherapy and at least 1 additional regimen for treatment of NSCLC
* World Health Organisation (WHO) Performance Status of 0 or 1
* Estimated life expectancy of more than 12 weeks
* Patient's tumour sample must be PD-L1 positive (≥25%of tumour cells with membrane staining (Cohort 1 and 2) or PD-L1 positive with ≥90% of tumour cells with membrane staining (Cohort 3))

Exclusion Criteria:

* Prior exposure to any anti-PD-1 or anti-PD-L1 antibody
* Brain metastases or spinal cord compression or unless asymptomatic, treated and stable (not requiring steroids).
* Active or prior autoimmune disease or history of immunodeficiency
* Evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses or active infections including hepatitis B, C and HIV.
* Evidence of uncontrolled illness such as symptomatic congestive heart failure, uncontrolled hypertension or unstable angina pectoris.
* Any unresolved toxicity CTCAE >Grade 2 from previous anti-cancer therapy.
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
* Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2025-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Dennis, MD, PhD, Study Director — AstraZeneca
Locations (117):
- United States (25):
  - Research Site, Goodyear, Arizona
  - Research Site, Santa Rosa, California
  - Research Site, New Haven, Connecticut
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Tampa, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, Waterloo, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Bethesda, Maryland
  - Research Site, Burlington, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Huntersville, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Fargo, North Dakota
  - Research Site, Blue Ash, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Spokane, Washington
  - Research Site, Wenatchee, Washington
- Research Site, Vienna, Austria
- Belgium (6):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Gilly
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
- Canada (5):
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Regina, Saskatchewan
- Czechia (2):
  - Research Site, Brno
  - Research Site, Prague
- France (10):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Marseille
  - Research Site, Pessac
  - Research Site, Rennes
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
- Germany (9):
  - Research Site, Berlin
  - Research Site, Borstel
  - Research Site, Cologne
  - Research Site, Dortmund
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Heidelberg
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Szolnok
  - Research Site, Tatabánya
  - Research Site, Törökbálint
- Italy (9):
  - Research Site, Candiolo
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Orbassano
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (21):
  - Research Site, Akashi-shi
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Habikino-shi
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Nagoya
  - Research Site, Natori-shi
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sayama
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Ube-shi
  - Research Site, Yokohama
- Philippines (2):
  - Research Site, Cebu City
  - Research Site, Quezon City
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Warsaw
- Research Site, Singapore, Singapore
- South Korea (4):
  - Research Site, Goyang-si
  - Research Site, Hwasun-gun
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (2):
  - Research Site, Hat Yai
  - Research Site, Muang
- United Kingdom (4):
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Gavrilov S, Zhudenkov K, Helmlinger G, Dunyak J, Peskov K, Aksenov S. Longitudinal Tumor Size and Neutrophil-to-Lymphocyte Ratio Are Prognostic Biomarkers for Overall Survival in Patients With Advanced Non-Small Cell Lung Cancer Treated With Durvalumab. CPT Pharmacometrics Syst Pharmacol. 2021 Jan;10(1):67-74. doi: 10.1002/psp4.12578. Epub 2020 Dec 21. PMID 33319498
- [Derived] Zhang Q, Luo J, Wu S, Si H, Gao C, Xu W, Abdullah SE, Higgs BW, Dennis PA, van der Heijden MS, Segal NH, Chaft JE, Hembrough T, Barrett JC, Hellmann MD. Prognostic and Predictive Impact of Circulating Tumor DNA in Patients with Advanced Cancers Treated with Immune Checkpoint Blockade. Cancer Discov. 2020 Dec;10(12):1842-1853. doi: 10.1158/2159-8290.CD-20-0047. Epub 2020 Aug 14. PMID 32816849
- [Derived] Garassino MC, Cho BC, Kim JH, Mazieres J, Vansteenkiste J, Lena H, Jaime JC, Gray JE, Powderly J, Chouaid C, Bidoli P, Wheatley-Price P, Park K, Soo RA, Poole L, Wadsworth C, Dennis PA, Rizvi NA. Final overall survival and safety update for durvalumab in third- or later-line advanced NSCLC: The phase II ATLANTIC study. Lung Cancer. 2020 Sep;147:137-142. doi: 10.1016/j.lungcan.2020.06.032. Epub 2020 Jun 30. PMID 32702570
- [Derived] Ouwens MJNM, Mukhopadhyay P, Zhang Y, Huang M, Latimer N, Briggs A. Estimating Lifetime Benefits Associated with Immuno-Oncology Therapies: Challenges and Approaches for Overall Survival Extrapolations. Pharmacoeconomics. 2019 Sep;37(9):1129-1138. doi: 10.1007/s40273-019-00806-4. PMID 31102143
- [Derived] Garassino MC, Cho BC, Kim JH, Mazieres J, Vansteenkiste J, Lena H, Corral Jaime J, Gray JE, Powderly J, Chouaid C, Bidoli P, Wheatley-Price P, Park K, Soo RA, Huang Y, Wadsworth C, Dennis PA, Rizvi NA; ATLANTIC Investigators. Durvalumab as third-line or later treatment for advanced non-small-cell lung cancer (ATLANTIC): an open-label, single-arm, phase 2 study. Lancet Oncol. 2018 Apr;19(4):521-536. doi: 10.1016/S1470-2045(18)30144-X. Epub 2018 Mar 12. PMID 29545095
- See also: AstraZeneca Cancer Study Locator Service astrazeneca@emergingmed.com 1-877-400-4656 — http://www.emergingmed.com
- See also: d4191c00003 revised csp 4 Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2583&filename=d4191c00003-revised-csp-4_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: 25 Feb 2014; Last patient in: 28 Dec 2015. Primary Analysis data cut-off (DCO): 03 Jun 2016; Final Analysis DCO: 7 Nov 2017. Patients were treated with durvalumab (10 milligrams [mg] / kilogram [kg] every 2 weeks [Q2W] intravenously [iv]). 101 sites in 16 countries treated patients in this study.
Pre-assignment Details: Patients were enrolled in 3 cohorts. Cohort enrolment was dependent upon epidermal growth factor receptor (EGFR) / anaplastic lymphoma kinase (ALK) status and programmed cell death ligand-1 (PD-L1) expression level (percent of tumor cells [TC] with membrane staining).
Groups:
- Cohort 1 (EGFR/ALK+): Consisted of patients who were EGFR/ALK positive and retrospectively or prospectively determined to be PD-L1 high (TC >=25%). In addition, the cohort included patients enrolled prior to Amendment 1 who were retrospectively determined to be PD-L1 low/neg (TC <25%) or PD-L1 status unknown.
- Cohort 2: Consisted of patients who were EGFR/ALK wild type/unknown and retrospectively or prospectively determined to be PD-L1 high (TC >=25%). In addition, the cohort included patients enrolled prior to Amendment 1 who were retrospectively determined to be PD-L1 low/neg (TC <25%) or PD-L1 status unknown.
- Cohort 3 (TC >= 90%): Consisted of patients who were EGFR/ALK wild type/unknown and prospectively determined to be PD-L1 high (TC >=90%).
Period: Overall Study
Arm/Group | Cohort 1 (EGFR/ALK+) | Cohort 2 | Cohort 3 (TC >= 90%)
Started | 111 (Treated) | 265 (Treated) | 68 (Treated)
Completed 12 Months of Treatment | 18 | 60 | 26
Completed | 0 | 0 | 0
Not Completed | 111 | 265 | 68
Not completed — Withdrawal by Subject | 20 | 20 | 3
Not completed — Death | 68 | 207 | 40
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Terminated from study at final DCO | 23 | 36 | 25

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on the safety analysis set, defined as all patients who received at least 1 dose of durvalumab and for whom any postdose data were available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (EGFR/ALK+) | Cohort 2 | Cohort 3 (TC >= 90%) | Total
Number analyzed (Participants) | 111 | 265 | 68 | 444
Age, Categorical [Count of Participants; unit: Participants] — age groups of <=18, between 18 and 65, >=65,
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 66 | 155 | 44 | 265
    >=65 years | 45 | 110 | 24 | 179
Age, Continuous [Median (Standard Deviation); unit: years] | 61.0 (11.45) | 62.0 (9.35) | 61.0 (10.58) | 62.0 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 103 | 29 | 202
  Male | 41 | 162 | 39 | 242
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 212 | 42 | 298
  Black or African American | 1 | 2 | 2 | 5
  Asian | 66 | 51 | 24 | 141
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 19 | 2 | 27
  Not Hispanic or Latino | 105 | 246 | 66 | 417
Weight [Median (Standard Deviation); unit: kg] | 59 (14.15) | 68 (14.52) | 66 (15.79) | 66 (14.93)
Weight group [Count of Participants; unit: Participants]
  <70 kg | 81 | 146 | 40 | 267
  Between 70 and 90 kg | 27 | 97 | 21 | 145
  >90 kg | 3 | 22 | 7 | 32
WHO performance status [Count of Participants; unit: Participants]
  (0) Normal activity | 45 | 86 | 19 | 150
  (1) Restricted activity | 65 | 178 | 49 | 292
  (2) In bed <=50% of the time | 1 | 1 | 0 | 2
  (3) In bed >50% of the time | 0 | 0 | 0 | 0
  (4) 100% bed ridden | 0 | 0 | 0 | 0
Primary tumor location [Count of Participants; unit: Participants] — Lung
  Participants | 111 | 265 | 68 | 444
Histology type [Count of Participants; unit: Participants]
  Squamous | 1 | 55 | 20 | 76
  Non-squamous | 110 | 210 | 48 | 368
AJCC staging at initial diagnosis [Count of Participants; unit: Participants] — Per tumor, node, metastasis (TNM) staging system as specified by American Joint Committee on Cancer (AJCC). The staging is determined by a number of different parameters and the higher the staging the worse the prognosis for survival.
  Participants
    Stage IA | 2 | 3 | 0 | 5
    Stage IB | 0 | 4 | 0 | 4
    Stage II | 0 | 1 | 0 | 1
    Stage IIA | 1 | 1 | 1 | 3
    Stage IIB | 0 | 5 | 0 | 5
    Stage III | 0 | 1 | 0 | 1
    Stage IIIA | 9 | 13 | 5 | 27
    Stage IIIB | 8 | 28 | 9 | 45
    Stage IV | 90 | 208 | 53 | 351
    Missing | 1 | 1 | 0 | 2
Best response to previous therapy [Count of Participants; unit: Participants] — based on the last therapy received prior to entering the study
  Participants
    complete response | 0 | 1 | 0 | 1
    partial response | 31 | 39 | 18 | 88
    stable disease | 34 | 86 | 18 | 138
    progression | 38 | 114 | 26 | 178
    non-evaluable | 2 | 15 | 2 | 19
    not applicable | 6 | 10 | 4 | 20
Time from informed consent to first dose [Count of Participants; unit: Participants]
  <=14 days | 21 | 68 | 7 | 96
  Between 14 and 21 days | 24 | 73 | 13 | 110
  between 21 and 42 days | 65 | 111 | 45 | 221
  > 42 days | 1 | 13 | 3 | 17
Overall disease classification [Count of Participants; unit: Participants] — either patient has any metastatic site of disease or has only locally advanced sites of disease
  Participants
    Metastatic | 102 | 245 | 61 | 408
    Locally advanced | 9 | 20 | 7 | 36
PD-L1 expression level [Number; unit: Number of patients (per PD-L1 category)] — % of tumor cells with membrane staining for PD-L1
  Number of patients (per PD-L1 category)
    Positive (>=25%) | 77 | 149 | 68 | 294
    Negative (<25%) | 30 | 95 | 0 | 125
    Positive (>=90%) | 47 | 72 | 67 | 186
    <90% | 33 | 122 | 0 | 155
    Unknown | 3 | 21 | 0 | 24
    Missing | 1 | 0 | 0 | 1
    Total per cohort | 111 | 265 | 68 | 444
Smoking history [Count of Participants; unit: Participants] — Patients who checked options Cigarettes, Cigarillos, Cigars, Pipe Tobacco, or Tobacco for Smoking are considered smokers.
  Participants
    Non-smoker | 65 | 39 | 9 | 113
    Smoker | 46 | 225 | 59 | 330
    Missing | 0 | 1 | 0 | 1
Number of regimens of previous anti-cancer therapy [Median (Standard Deviation); unit: Number of regimens] | 3 (2.00) | 3 (1.38) | 2 (0.80) | 3 (1.54)

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Patients commenced treatment with durvalumab on Day 1 and continued on a Q2W schedule for a maximum of 12 months. Tumor assessments using computed tomography / magnetic resonance imaging were performed every 8 weeks. Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) measurements as given by the Independent Central Review (ICR) were used to derive the primary variable of ORR .
Time Frame: Responses recorded during initial 12 month treatment period (up to primary analysis DCO)
Population: The "Full analysis set [FAS] - evaluable for response per ICR" set, included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the ICR.
Measure: Number (95% Confidence Interval); unit: % of patients evaluable for response
Groups:
- Cohort 1 (EGFR/ALK+) PD-L1+ (>=25%): Consisted of patients who were EGFR/ALK positive and retrospectively or prospectively determined to be PD-L1 high (TC >=25%). In addition, the cohort included patients enrolled prior to Amendment 1 who were retrospectively determined to be PD-L1 low/neg (TC <25%) or PD-L1 status unknown. patients with PD-L1 TC>=90% are included in this group.
- Cohort 1 (EGFR/ALK+) PD-L1+ (<25%): Consisted of patients who were EGFR/ALK positive and retrospectively or prospectively determined to be PD-L1 high (TC >=25%). In addition, the cohort included patients enrolled prior to Amendment 1 who were retrospectively determined to be PD-L1 low/neg (TC <25%) or PD-L1 status unknown.
- Cohort 2 PD-L1+ (>=25%): Consisted of patients who were EGFR/ALK wild type/unknown and retrospectively or prospectively determined to be PD-L1 high (TC >=25%). In addition, the cohort included patients enrolled prior to Amendment 1 who were retrospectively determined to be PD-L1 low/neg (TC <25%) or PD-L1 status unknown. Patients with PD-L1 TC>=90% are included within the PD-L1 high (TC>=25%) group.
- Cohort 2 PD-L1+ (<25%): Consisted of patients who were EGFR/ALK wild type/unknown and retrospectively or prospectively determined to be PD-L1 high (TC >=25%). In addition, the cohort included patients enrolled prior to Amendment 1 who were retrospectively determined to be PD-L1 low/neg (TC <25%) or PD-L1 status unknown.
- Cohort 3 (TC>=90%): Consisted of patients who were EGFR/ALK wild type/unknown and prospectively determined to be PD-L1 high (TC>=90%).
Arm/Group | Cohort 1 (EGFR/ALK+) PD-L1+ (>=25%) | Cohort 1 (EGFR/ALK+) PD-L1+ (<25%) | Cohort 2 PD-L1+ (>=25%) | Cohort 2 PD-L1+ (<25%) | Cohort 3 (TC>=90%)
Number analyzed (Participants) | 74 | 28 | 146 | 93 | 68
% of patients evaluable for response | 12.2 [5.7 to 21.8] | 3.6 [0.1 to 18.3] | 16.4 [10.8 to 23.5] | 7.5 [3.1 to 14.9] | 30.9 [20.2 to 43.3]

2. Secondary Outcome: Time to Response (TTR)
Description: TTR (per RECIST 1.1 as assessed by the ICR) is defined as the time from the date of first dose until the date of first documented response (which is subsequently confirmed). TTR was only analyzed for Cohort 2.
Time Frame: Responses recorded during initial 12 month treatment period (up to primary analysis DCO)
Population: The "FAS - evaluable for response per ICR" set for Cohort 2, included all treated patients in Cohort 2 who had a baseline tumor assessment and had measurable disease at baseline according to the ICR.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 (EGFR/ALK+) PD-L1+ (>=25%) | Cohort 1 (EGFR/ALK+) PD-L1+ (<25%) | Cohort 2 PD-L1+ (>=25%) | Cohort 2 PD-L1+ (<25%) | Cohort 3 (TC>=90%)
Number analyzed (Participants) | 0 | 0 | 24 | 7 | 0
Months |  |  | 1.9 [1.6 to 16.7] | 2.1 [1.7 to 13.8] |

3. Secondary Outcome: Duration of Response (DoR)
Description: DoR (per RECIST 1.1 as assessed by the ICR) was defined as the time from the date of first documented response (which was subsequently confirmed) until the first date of documented progression or death in the absence of disease progression (ie, date of PFS event or censoring - date of first response + 1). DoR was only analyzed for Cohort 2. Cohort 2: Median DoR was 12.3 months in the PD-L1 high (TC>=25%) group at DCO (Q3 was NR). Of the 7 evaluable patients, the median DoR was not reached in the PD-L1 low/neg group (TC <25%); therefore the DoR "number of participants analyzed" field has been entered as "0" and the DoR results field has been left blank.
Time Frame: Time from response to progression, death, or last assessment (up to approximately 2 years 3 months for the primary analysis DCO)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort 1 (EGFR/ALK+) PD-L1+ (>=25%) | Cohort 1 (EGFR/ALK+) PD-L1+ (<25%) | Cohort 2 PD-L1+ (>=25%) | Cohort 2 PD-L1+ (<25%) | Cohort 3 (TC>=90%)
Number analyzed (Participants) | 0 | 0 | 24 | 0 | 0
Months |  |  | 12.3 [7.5 to NA] — 75th percentile not reached (NR) |  |

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose until death due to any cause (ie, date of death or censoring - date of first dose + 1). Results are reported as median OS, calculated using the Kaplan-Meier methodology.
Time Frame: From date of first treatment until final DCO (up to approximately 3 years 8 months)
Population: The FAS included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (EGFR/ALK+) PD-L1+ (>=25%) | Cohort 1 (EGFR/ALK+) PD-L1+ (<25%) | Cohort 2 PD-L1+ (>=25%) | Cohort 2 PD-L1+ (<25%) | Cohort 3 (TC>=90%)
Number analyzed (Participants) | 77 | 30 | 149 | 94 | 67
Months | 13.3 [6.3 to 24.5] | 9.9 [4.2 to 13.3] | 10.9 [8.6 to 13.6] | 9.3 [5.9 to 10.8] | 13.2 [5.9 to NA] — The upper limit of 95% confidence interval was not reached for patients in Cohort 3.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) observed up until 90 days following discontinuation of durvalumab or until the initiation of the first subsequent anticancer therapy following discontinuation of durvalumab (whichever occurred first).
Description: All-Cause Mortality is reported for the overall study period, up to the final DCO. Serious and Other (non-serious) TEAE data is reported for the initial treatment phase (maximum of 12 months of treatment).
Groups:
- Cohort 3 (TC >=90%): Consisted of patients who were EGFR/ALK wild type/unknown and prospectively determined to be PD-L1 high (TC >=90%).
Arm/Group | Cohort 1 (EGFR/ALK+) | Cohort 2 | Cohort 3 (TC >=90%)
All-Cause Mortality (participants affected / at risk) | 70/111 | 217/265 | 41/68
Serious Adverse Events (participants affected / at risk) | 18/111 | 77/265 | 24/68
Other Adverse Events (participants affected / at risk) | 96/111 | 233/265 | 60/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (EGFR/ALK+) (N=111) | Cohort 2 (N=265) | Cohort 3 (TC >=90%) (N=68)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (7) | 2 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (3) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic atrophy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 8 (9) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Central nervous system infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (EGFR/ALK+) (N=111) | Cohort 2 (N=265) | Cohort 3 (TC >=90%) (N=68)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 43 (52) | 8 (8)
Hyperthyroidism (Endocrine disorders) | 11 (12) | 17 (18) | 7 (8)
Hypothyroidism (Endocrine disorders) | 11 (14) | 19 (24) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 10 (10) | 4 (6)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8) | 12 (12) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (15) | 37 (45) | 16 (19)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 39 (53) | 9 (10)
Nausea (Gastrointestinal disorders) | 14 (16) | 46 (57) | 12 (15)
Vomiting (Gastrointestinal disorders) | 13 (15) | 27 (36) | 10 (13)
Asthenia (General disorders) | 14 (15) | 53 (76) | 4 (4)
Fatigue (General disorders) | 15 (16) | 69 (80) | 20 (31)
Non-cardiac chest pain (General disorders) | 3 (4) | 10 (15) | 4 (5)
Oedema peripheral (General disorders) | 7 (8) | 25 (25) | 9 (13)
Pain (General disorders) | 1 (1) | 8 (8) | 4 (4)
Pyrexia (General disorders) | 12 (14) | 53 (81) | 12 (16)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 6 (9) | 8 (8) | 6 (6)
Urinary tract infection (Infections and infestations) | 4 (4) | 15 (19) | 3 (4)
Viral upper respiratory tract infection (Infections and infestations) | 5 (6) | 12 (13) | 11 (18)
Alanine aminotransferase increased (Investigations) | 5 (5) | 11 (13) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 12 (14) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 14 (14) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 15 (15) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 22 (22) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15) | 71 (77) | 12 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 14 (20) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 21 (25) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 23 (24) | 8 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 16 (21) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 18 (21) | 2 (2)
Dizziness (Nervous system disorders) | 6 (6) | 12 (18) | 4 (6)
Headache (Nervous system disorders) | 13 (15) | 26 (32) | 6 (6)
Anxiety (Psychiatric disorders) | 2 (2) | 16 (16) | 2 (2)
Insomnia (Psychiatric disorders) | 10 (12) | 16 (19) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (32) | 56 (67) | 13 (16)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 14 (15) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 43 (46) | 7 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 14 (20) | 4 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 20 (23) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (11) | 27 (39) | 13 (14)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 19 (20) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No